CLINICAL TRIAL: NCT00361023
Title: Effects of Angiotensin Type 1 Receptor Blockade With Losartan on Insulin Sensitivity and Secretion in Subjects With Type 2 Diabetes and Nephropathy
Brief Title: Effects of Losartan on Insulin Sensitivity and Secretion in Type 2 Diabetes and Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LISS
Record Dates: First submitted 2006-08-01; First posted 2006-08-07 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-01

CONDITIONS: Type 2 Diabetes; Diabetic Nephropathy
Keywords: Angiotensin type 1 receptor blocker (ARB); losartan; type 2 diabetes; insulin sensitivity and secretion; glucose metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Insulin Resistance | interventions — Losartan

INTERVENTIONS:
Drug: losartan

SUMMARY:
Angiotensin type-1 receptor (AT1R) blockers (ARBs) have been recognized recently as regulators of glucose and lipid metabolism in adipocytes and adipose tissue.Moreover telmisartan and irbesartan have been recognized recently as regulators of glucose metabolism. For ARB losartan, the results were controversial. To confirm its effect on glucose metabolism, we designed and performed a prospective, randomized and controlled study in subjects with type 2 diabetes and nephropathy.

DETAILED DESCRIPTION:
Angiotensin II (AngII), the main effector peptide of the rennin-angiotensin system (RAS), is implicated in the development of vascular, cardiac, and renal pathologies. Several lines of evidence have suggested that AngII can impair insulin sensitivity.Angiotensin type-1 receptor (AT1R) blockers (ARBs) have been recognized recently as regulators of glucose and lipid metabolism in adipocytes and adipose tissue. Recent clinical trials suggest that blockade of the RAS, either by inhibiting the angiotensin-converting enzyme (ACE) or by blocking AT1R, may substantially lower the risk for type 2 diabetes. In the Heart Outcomes Prevention Evaluation (HOPE) trial, there was 34% reduction in relative risk for the development of type 2 diabetes. Similarly, in the Intervention For Endpoint Reduction in Hypertension study (LIFE), the incidence of type 2 diabetes was reduced by 25% in the losartan group compared with other antihypertensive therapies. Previous study demonstrated that AT1R blockade improved insulin sensitivity in animal models of insulin resistance. The underlying mechanism of the insulin sensitizing and anti-diabetic effect of ARBs is incompletely clear.

The nuclear hormone receptor peroxisome proliferator activated receptor- (PPAR-γ) plays an important role in the regulation of insulin sensitivity. Several studies have shown the ARBs telmisartan and irbesartan potently induces PPAR-γ activity, promoting PPAR-γ-dependent differentiation in adipocytes. However, not all ARBs own PPAR-γ activating properties. In vitro studies have shown that significant differences among PPAR-γ activating ARBs are likely caused by their physicochemical properties, and high lipophilicity is required to obtain sufficiently high penetration rates to bind to intracellular PPAR-γ. Losartan at high concentrations could activate PPAR-γ and behaved like partial PPAR-γ agonists. Nevertheless the results of losartan on insulin sensitivity remain controversial.

To elucidate the underlying effects of losartan on insulin sensitivity, we investigated the effects of losartan on insulin sensitivity and secretion in patients with type 2 diabetes and nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose (FPG) level of 3.3-9.0mmol/L
* 2h plasma glucose level of 7.5-13 mmol/L
* Body mass index (BMI) of 22 kg/m2
* Two occasions of a ratio of urinary albumin to urinary creatinine≥300 or 24 hours urinary protein concentration is >150mg.
* Informed consent

Exclusion Criteria:

* Type1 diabetes or nondiabetic renal disease

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2006-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Hui M Jin, MD, Principal Investigator — Shanghai NO.3 people's Hospital